CLINICAL TRIAL: NCT02213718
Title: The Effect of Desflurane on Myocardial Function in Patients Undergoing Coronary Artery Bypass Grafting
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xin Chen, staff, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20140607; 20140627 (Other: the ethic committee of tongji hospital)
Record Dates: First submitted 2014-07-31; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Bypass Graft Redo; General Anesthetic Drug Adverse Reaction
Keywords: Desflurane; myocardial function; Coronary Artery Bypass Surgery
MeSH Terms: interventions — Desflurane; Propofol; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desflurane (Experimental): desflurane (7%-8% end-tidal concentration), sufentanil (TCI: 2-3 ng/ml) and vecuronium (0.04mg/kg/h)
  Interventions: Drug: Desflurane; Drug: sufentanil
- propofol (Active Comparator): intravenous administration of sufentanil (1μg/kg), etomidate(0.3mg/kg) and vecuronium (0.08mg/kg). The anesthesia is maintained with propofol (TCI:3.5-4.0μg/min), sufentanil (TCI: 2-3 ng/ml) and vecuronium (0.04mg/kg/h).
  Interventions: Drug: propofol; Drug: sufentanil

INTERVENTIONS:
Drug: Desflurane — desflurane (7%-8% end-tidal concentration)
  Other Names: brand names：Baxter; serial numbers and code names：not available yet
  Arms: Desflurane
Drug: propofol — propofol (TCI:3.5-4.0μg/min)
  Other Names: brand name：Diprivan; serial numbers and code names：not available yet
  Arms: propofol
Drug: sufentanil — TCI: 2-3 ng/ml during the duration of surgery, an expected average of 4 hours
  Other Names: brand name: Yichang Humanwell pharmaceutical co.,LTD; serial numbers and code names: not available yet

SUMMARY:
This study is to assess the effect of desflurane on myocardial function in patents who underwent coronary artery bypass grafting.

DETAILED DESCRIPTION:
Desﬂurane, one of the third-generation inhaled anesthetics, is introduced in clinical practice in 1990s. Decades of clinical use has provided evidence for desﬂurane's safe and efﬁcacious use as a general anesthetic. Compared with other volatile anesthestics, it has several characteristics: lower blood and lipid solubility, more stable in vitro and the lowest in vivo metabolism. Its particular low fat solubility properties promote rapid equilibration and rapid elimination at the end of anesthesia which reduces slow compartment accumulation and promotes predictable emergence, early extubation, and the ability to rapidly transfer patients from the operating room to the recovery unit. In addition, several investigations found that patients with desflurane anesthesia recovered their protective airway reﬂexes and awakened to a degree sufﬁcient to minimize the stay in the high dependency recovery area.

A burgeoning body of investigations has shown that desflurane can directly act on myocardial and vascular functions. Desflurane has coronary vasodilative effects in in situ canine hearts which is comparable to sevoflurane does. Although it is controversial regarding to the effect of desflurane on myocardial excitation-contraction coupling and electrophysiologic behavior, a elaborated study found desflurane induced a positive inotropic effect in rat myocardium in vitro compared with isoflurane. A recent study suggested that desflurane decreased right ventricular contractility much less and maintained the right over left pressures ratio at more favorable values compared with sevoflurane. Furthermore, substantial investigations found that clinically relevant concentration desflurane preconditioning or postconditioning could protect myocardium from ischemia-reperfusion in mammalian animal models or isolated human cardiac tissues. However, it is unclear whether desflurane can provide protection for patients with coronary artery disease. Therefore, this study is designed to investigate the effect of desflurane on myocardial function in patents who underwent coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CAD 2. ASAⅡ～Ⅲ

-

Exclusion Criteria:

1. Left ventricular ejection fraction <40%
2. Left ventricular aneurysm
3. Acute myocardial infarction in latest two weeks, atrial fibrillation
4. Associated vascular diseases, severe systemic diseases involving the renal and hepatic systems
5. Respiratory disease( forced vital capacity less than 50% of predicted values )
6. Preoperative left bundle branch block -

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Serum Concentration of cTnI | 48 hours
  at the begingineg of the surgery,immediately after surgery,4 hours after the surgery, 8 hours after the surgery, 12 hours after the surgery, 24 hours after the surgery

SECONDARY OUTCOMES:
Continuous Monitoring of ECG | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  participants will be followed for the duration of hospital stay, an expected average of 5 weeks.ECG incidents such as tachycardia, bradycardia, premature ventricualr contraction and ST segment changes will be monitored and recorded.

OTHER OUTCOMES:
Incidence of segmental wall motion | Incidence of segmental wall motions will be monitored during the surgery, an expected average of 4 hours.
  Incidence of segmental wall motions will be monitored during the surgery, an expected average of 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ailin Luo, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Dept. of Anesthesiolgy, Tongji hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- See also: educational — http://www.hust.edu.cn/
- See also: educational — http://www.tjmu.edu.cn/
- See also: research — http://www.tjh.com.cn/